CLINICAL TRIAL: NCT01848652
Title: Phase II Study Evaluating the Combination Pegylated Liposomal Doxorubicin and Dexamethasone for the Treatment of Immunocompetent Patients With Cerebral Lymphoma Relapsed or Refractory to First-line Chemotherapy Containing High Dose Methotrexate (MTXHD) and / or High-dose Cytarabine.
Brief Title: Phase II Study Evaluating a Combination of Pegylated Liposomal Doxorubicin and Dexamethasone for the Treatment of Immunocompetent Patients With Cerebral Lymphoma Relapsed or Refractory to First-line Chemotherapy With High Dose Methotrexate (MTXHD) and / or High-dose Cytarabine.
Acronym: MYLY
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The laboratory's partner on this study decides to terminate the contract with the CHRU Brest, because of the difficulty of the recruitment.
Sponsor: University Hospital, Brest (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RB 12.032 - MYLY
Record Dates: First submitted 2013-05-03; First posted 2013-05-07 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Cerebral Lymphoma B Cell Refractory
Keywords: cerebral lymphoma B cell refractory; Myocet; efficacy; safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MYOCET (Experimental)
  Interventions: Drug: infusion of MYOCET

INTERVENTIONS:
Drug: infusion of MYOCET

SUMMARY:
The protocol is to assess the overall response rate (complete response and partial response) of treatment with non-pegylated liposomal doxorubicin at a dose of 50 mg / m² in combination with dexamethasone in immunocompetent adult patients with primary brain lymphoma large B-cell refractory or relapsed after first-line treatment MTXHD and high-dose cytarabine, excluding strict eye lymphomas.

This is a Phase II, open, prospective, multicenter, non-comparative with direct individual benefit.

ELIGIBILITY:
Inclusion Criteria:

* Patient with cerebral lymphoma B cell refractory or relapsed within 12 months after first-line chemotherapy with high-dose methotrexate (1.5 g / m²) and high dose cytarabine (2g / m²) and / or radiotherapy or autologous, or patient with an indication against these treatments.

Refractory disease is defined by the absence of objective response to treatment or relapse within 3 months of it. A relapse is defined as disease progression after obtaining a complete or partial response.

* Age greater than or equal to 18 years
* Performance Index less than 4
* Illness measured by CT or MRI
* Hematologic adequate: neutrophils> 1.5 x 106 / L, platelets> 100x106 / L
* Adequate hepatic function: ALT / AST and bilirubin less than the upper limit of the normal laboratory
* Adequate renal function: creatinine clearance greater than 60 ml / min
* adequate cardiac function measured by ejection fraction of the left ventricle> 50% by echocardiography
* Informed consent signed
* Negative pregnancy test for women of childbearing age
* Able to understand the arrangements for monitoring the study and to comply
* Corticosteroids are only accepted during the first cycle

Exclusion Criteria:

* Patients with immunosuppression from any cause (HIV, history of transplantation, immunosuppressive treatments ...)
* Prior treatment MYOCET ® or other anthracycline
* Active infection
* Surgery large (more than 3 days hospitalization) within 28 days before enrollment in the study, except for a diagnostic neurosurgical
* Hypersensitivity to any component of the treatment
* Contraindications to the administration of MYOCET ® and / or dexamethasone Participation in a clinical trial within 4 weeks prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Answer at treatment | after 2 cycles of treatment (84 days)
  Answer, whether complete or partial, according to the International Primary CNS Lymphoma Collaborative Group (IPCG) (ASH 2004) after two cycles of treatment (4 infusions MYOCET ®).

SECONDARY OUTCOMES:
Tolerance at treatment | after each cycle and until the end of follow
  Tolerance, assessed according to the criteria of the National Cancer Institute (NCI)-Common Toxicity Criteria (CTC) version (version 4.03) after administration of each cycle, overall survival, progression-free and disease-free event for complete responses.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian TEMPESCUL, Dr, Principal Investigator — University hospital of Brest
Locations (3):
- France (3):
  - CHRU de Brest, Brest
  - Hôpital Pitié Salpêtrière, Paris
  - CHU de Rennes Hôpital Pontchaillou, Rennes